CLINICAL TRIAL: NCT00163956
Title: Failed Retrieval of Inferior Vena Cava (IVC) Filters: Long-Term Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Other Study IDs: AlfRad2005-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-09

CONDITIONS: DVT; PE
Keywords: IVC filters; failed retrieval

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The inferior vena cava (IVC) is a large vein that enters the bottom part of the heart. Venous blood from the lower portion of the body drains into the IVC. The IVC then returns blood back to the heart. An IVC filter is placed to help prevent the blood clots moving from the legs to the heart or lung. The idea behind using a filter in the IVC is to capture potential fatal pulmonary emboli at an anatomical location where they may pose less risk for the patient. Early filters, 1960's and 70's were, remained in the vein permanently. More recently, temporary or retrievable filters have been developed and are being widely used.

Complications have been demonstrated with long-term placement of IVC filters. In a randomised study it was found that that patients with IVC filter placement had greater than three times the incidence of recurrent deep vein thrombosis (DVT) compared to their control population at two years. Blockage of the vein, recurrent pulmonary emboli, filter penetration and filter fragmentation have all been described.

With the advent of retrievable filters (filters that can be place temporarily and then removed at a later date) there has been renewed popularity for placement of temporary filters. To our knowledge, no one has yet to follow the population of intended temporary IVC filters, who undergo failed retrieval, and consequently end up with a permanent IVC filter.

We plan to prospectively enrol 40 Alfred patients who have undergone a temporary IVC filter placement and subsequently have had failed IVC filter retrieval.

Our aim is to evaluate the long term outcomes for patients with failed IVC retrieval.

Specifically we will determine the risk, due to failed filter retrieval, of:

* IVC stenosis
* IVC occlusion
* Development of DVT and
* analyse the clinical outcomes (symptoms), their prevalence and their distribution

Patients will receive routine care and their data will be analysed annually as collected. The follow-up period is indefinite and will be at the discretion of the treating doctor.

DETAILED DESCRIPTION:
Clinical Study Protocol

Failed Retrieval of Inferior Vena Cava (IVC) filters: long-term outcomes

Study Objective To evaluate the long term outcomes for failed IVC retrieval.

Background Long-term placement of IVC filters is not without complication. Descosous et al. demonstrated that those patients with IVC filter placement had greater than three times the incidence of recurrent DVT at two years. Pulmonary Emboli (PE) have been reported. These can occur when there is no evidence of PE prior to insertion of the IVC filter. This was shown by Rogers et al where 2.3% of trauma patients receiving prophylactic filters developed a PE. They can also occur as a recurrence (i.e. where a PE has already been demonstrated prior IVC filter insertion) in 2.5 to 7.7 % of patients1, 2.

Caval thrombosis resulting in occlusion have been reported to occur in between 1-24% of cases depending on the type of filter3, 4. Guidewire and catheter entrapment during central venous and pulmonary artery catheter placement have also been reported as long term IVC filters become more prevalent. Filter penetration and filter fragmentation have all been described.

With the advent of retrievable filters there is renewed popularity for temporary caval interruption. To our knowledge, no one has yet to follow the population of intended temporary caval interruption, who undergo failed retrieval, and consequently end up with a permanent IVC filter. This study will look at the incidence and degree of caval occlusion, caval stenosis and incidence of DVT in patients at The Alfred who have had a failed retrieval of an implanted IVC filter. Patient will be recruited for up to four years, the incidence of failed retrieval at The Alfred is 10 per year, and follow up will be ongoing.

Patient Population Alfred patients undergoing temporary IVC filter placement and subsequently have had failed IVC filter retrieval.

Study Design This is a prospective, single-arm study.

* Patients identified with failed filter retrieval will be asked to participate in the study. They will have a CT cavagram and lower limb duplex doppler ultrasound annually which is part of standard patient management practice.
* Clinical evaluation, history-taking and examination for filter complications and venous hypertension will be conducted annually, again as part of standard patient management.
* Data will be collected as per data collection forms and analysed.

Enrolment Size 40 patients will be enrolled.

Primary End-Points CT cavagram will be used to evaluate/measure:

* Caval occlusion.
* Caval stenosis.

Chronic or acute DVT will be evaluated with:

 Duplex sonography.

Secondary End-points Adverse events related to IVC filter as established through:

* Physical examination.
* Patient interview.

Research Plan

Specific Aim:

To evaluate the long term outcomes for failed IVC retrieval.

Objectives:

* To determine the risk of IVC stenosis due to failed filter retrieval.
* To determine the risk of IVC occlusion due to failed filter retrieval.
* To identify the risk of DVT due to failed filter retrieval.
* To analyse the clinical outcomes (symptoms), their prevalence and their distribution, produced as a result of failed filter retrieval.

Research Design and Methods:

This is a prospective, single-arm clinical study. An will be made to the HREC to obtain ethics approval for this study. Participants will be enrolled consecutively.

Patients will receive routine care and their data will be analysed annually as collected. The follow-up period is indefinite and will be at the discretion of the treating doctor.

The data from the CT cavagram and duplex Doppler will be collected by the research assistant from the patient's histories and reported onto the 'Investigations' data sheet (see Appendix I.)

The data from the clinical interview and examination will be collected from the patient's histories and reported onto the 'Examination' data sheet (see Appendix II.)

Analysis Plan and Statistical Methods:

This study will look at the incidence and degree of caval occlusion, caval stenosis and incidence of DVT in patients at The Alfred who have had a failed retrieval of an implanted IVC filter.

Data management, quality control Non-identifiable information will be collected and securely stored in the Radiology Department research office. Data will be entered into an excel spreadsheet and the incidence of the primary and secondary endpoints summarised.

Complications and Reporting of Adverse Events:

There are no direct medical complications that might arise due to participation in this trial as patients will have routine care. This study involves data collection and no change to routine management. Any adverse event in reporting identifiable data will be reported to the HREC committee within 24 hours from the identification of the event.

Complications resulting from the CT cavagram include:

* Contrast Allergy
* Anaphylaxis
* Infection

Adverse events therefore relate principally to confidentiality. See 'Data Management' below for procedures related to adverse event reporting for breach of confidentiality.

Data Management:

* Data will be collated, stored and analysed by the research coordinator, Dr. Helen Kavnoudias.
* All data forms will be de-identified prior to reporting and/or publication of results.
* Patient medical records will be appropriately labelled as participants of research study and kept indefinitely.
* All departmental procedures relating to research, ethics and privacy regulations will be adhered to.
* Adverse events involving data management will be reported to the ethics committee with 24-hours by the research team.

Time-frame:

This research will be ongoing. There are approximately 10 failed retrievals each year.

References:

1. Wolf F, Thurnher S, Lammer J (Simon nitinol vena cava filters: Effectiveness and complications) Rofo Fortschr Geb Rontgenstr Neuen Bildgeb Verfahr 2001; 173: 924-30.
2. Harries SR, Wells IP, Roobottom VA. Long term follow up of the antheor interior vena cava filter. Clin Radiol 1998; 53: 350-2
3. Millward SF, Peterson RA, Moher D, et al. LGM (Vena Tech) vena caval filter: Experience at a single institution. J Vase Interv Radiol 1994; 5:351-6.
4. Greenfield LJ, Proctor MC, Cho KJ, et al. Extended evaluations of the titanium Greenfield vena caval filter. J Vasc Surg 1996; 20: 458-65

Appendix I

Investigations

Date Follow-Up

Name

Sex

Age

UR

CT Cavagram Is there occlusion of the IVC? Yes No Is there >50% stenosis of the IVC? Yes No

Is there >20% stenosis of the IVC? Yes No

Duplex Doppler Is there presence of thrombus? Yes No

If yes, where?

Is the thrombus: Acute? Chronic?

Appendix II

Examination

Date Follow-Up

Name

Sex

Age

UR

Does the patient suffer from any of the following:

(please tick) ٱLower limb venous incompetence ٱ Chronic limb pain ٱ Oedema ٱ Discolouration ٱ Ulceration ٱ Historical episodes of DVT ٱ PE ٱ Filter-fragmentation embolisation

CEAP Score:

ELIGIBILITY:
Inclusion Criteria:

* na

Exclusion Criteria:

* na

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-08; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lyon, MBBS RANZCR, Principal Investigator — Bayside Health
Locations (1):
- Radiology Department, The Alfred, Melbourne, Victoria, Australia